CLINICAL TRIAL: NCT04388475
Title: A Phase II Open-label Study Investigating the Efficacy, Safety and Pharmacokinetic Properties of OKN-007 Combined With Temozolomide in Patients With Recurrent Glioblastoma
Brief Title: Open-label Study Investigating of OKN-007 Combined With Temozolomide in Patients With Recurrent Glioblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Oblato, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OKN-007-IV-RMG-201
Record Dates: First submitted 2020-05-06; First posted 2020-05-14 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Recurrent Malignant Glioma; Brain Glioblastoma
MeSH Terms: conditions — Glioma | interventions — OKN 007; disufenton sodium; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- All patients (Experimental): All patients enrolled in this study
  Interventions: Drug: OKN-007; Drug: Temozolomide (TMZ)

INTERVENTIONS:
Drug: OKN-007 — Drug: OKN-007 (400 mg OKN-007/mL in a phosphate buffer) Administered via IV infusion, at a dose level of 60 mg/kg, given three times a week for 12 weeks, two times a week for a further 12 weeks and once per week until disease progression or up to two years.
  Other Names: NXY-059, HPN-07
Drug: Temozolomide (TMZ) — Administered via oral, at a dose level of 150 mg/m2, once daily on Days 1-5 of each 28 day cycle in Cycle 1. If this dose level is tolerated, then in Cycle 2 (and subsequent cycles), at a dose level of 200 mg/m2, once daily on Days 1-5 of each 28 day cycle.
  Other Names: Temodar

SUMMARY:
This is a phase II open-label study investigating the efficacy, safety and pharmacokinetic(PK) properties of OKN-007 combined with temozolomide(TMZ) in patients with recurrent glioblastoma(GBM). All patients will have been previously treated with the standard-of-care treatment which includes surgical resection, radiation and chemotherapy, and in some cases treatment for recurrent disease. Patients with unequivocal recurrence (first or greater) established by MRI and meeting inclusion and exclusion criteria, will be eligible for OKN-007 treatment on this protocol.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed Glioblastoma based on histopathology or molecular profile analysis (WHO Grade IV), following primary treatment with TMZ and radiotherapy (minimum of 50 Gy) and at least two cycles of maintenance TMZ (5 days of a 28 day cycle) as first-line or second-line treatment with another treatment regimen, excluding bevacizumab.
2. Patients must have medical records available documenting O6-methylguanine-DNA methyltransferase (MGMT) promoter methylation status analysis or must have tumor tissue samples available from prior GBM surgery or open biopsy for MGMT status determination.
3. For patients with unresected recurrent tumor, unequivocal radiographic evidence of tumor progression by MRI. These patients must have at least one measurable lesion.
4. Patients with recent resection of recurrent viable tumor are eligible following post-operative MRI perfusion scan with or without measurable lesions.
5. No more than two prior lines of therapy for glioblastoma. Any second-line therapy is acceptable, excluding bevacizumab as second line.
6. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
7. Full recovery (≤ grade 1) from the toxic effects.
8. Adequate renal, liver and bone marrow function:

   * Hemoglobin >9.0 g/dL
   * Leukocytes >3,000/mcL
   * Absolute neutrophil count >1,500/mcL
   * Platelets >100,000/mcL
   * Total bilirubin ≤ 1.5 × upper limit of normal (ULN)
   * AST (SGOT) / ALT (SGPT) ≤2.5 × ULN
   * Creatinine clearance ≥ 60 mL/min
9. Patients must be ≥18 years of age

Exclusion Criteria:

1. Early discontinuation of TMZ in prior line due to treatment related Adverse events (AEs).
2. Second primary malignancy expected to require treatment within a 6 month period (except adequately treated basal cell carcinoma of the skin).
3. Have received treatment within the last 28 days with a drug that has not received regulatory approval for any indication at the time of study entry.
4. Have received chemotherapeutic agents (including temozolomide) within 28 days or within 5 half-lives for non-cytotoxic agents (whichever is shorter) of study entry
5. Serious concomitant systemic disorders
6. Patients with abnormal sodium, potassium, or creatinine levels ≥ grade 2.
7. Patients with prothrombin time/partial thromboplastin time (PT/PTT) or International normalized ratio (INR) above the ULN.
8. Inability to comply with protocol or study procedures.
9. Patients who have received bevacizumab for recurrent glioblastoma or are planning to initiate treatment with bevacizumab for tumor necrosis. (Past treatment with bevacizumab for tumor necrosis is acceptable).
10. Patients receiving or planning to initiate treatment with the tumor treating fields device (Optune®) (Optune® prior to enrollment is permitted).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-06-12 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
Incidents of Adverse Events during the subjects are taking OKN-007 with Temozolomide | Through study completion up to 24 months
  Evaluate incidents of Adverse Events during the subjects are taking OKN-007 with Temozolomide. Adverse events will be graded according to Common Terminology Criteria for Adverse Events (CTCAE, version 5.0).
Overall Survival (OS) rate | 6 months
  Proportion of subjects who are alive after six months of starting treatment. OS is defined as the time from first treatment dose until date of death due to any cause.

SECONDARY OUTCOMES:
Overall Response Rate (ORR%) | 24 months
  The proportion of patients with a complete response or partial response to treatment.
Progression Free Survival (PFS) rate | 6 months
  Proportion of subjects who are alive and progression free after six months of starting treatment. PFS is defined as the time from first treatment dose until objective tumor progression on the RANO criteria or death.
Cmax of OKN-007 in blood plasma | Day 1 and Day 5 in Cycle 1 and 2 (28 Day Cycle)
  The sample will be collected at 10 time points during 24 hours after OKN-007 administration.
AUC of OKN-007 in blood plasma | Day 1 and Day 5 in Cycle 1 and 2 (28 Day Cycle)
  The sample will be collected at 10 time points during 24 hours after OKN-007 administration.
Tmax of OKN-007 in blood plasma | Day 1 and Day 5 in Cycle 1 and 2 (28 Day Cycle)
  The sample will be collected at 10 time points during 24 hours after OKN-007 administration.
Cmax of Temozolomide in blood plasma | Day 1 and Day 5 in Cycle 1 and 2 (28 Day Cycle)
  The sample will be collected at 8 time points during 24 hours after Temozolomide administration.
AUC of Temozolomide in blood plasma | Day 1 and Day 5 in Cycle 1 and 2 (28 Day Cycle)
  The sample will be collected at 8 time points during 24 hours after Temozolomide administration.
Tmax of Temozolomide in blood plasma | Day 1 and Day 5 in Cycle 1 and 2 (28 Day Cycle)
  The sample will be collected at 8 time points during 24 hours after Temozolomide administration.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Providence Saint John's Health Center - John Wayne Cancer Institute, Santa Monica, California
  - Swedish Medical Center, Englewood, Colorado
  - AdventHealth Orlando, Orlando, Florida
  - University of Iowa, Iowa City, Iowa
  - Norton Healthcare, Louisville, Kentucky
  - Henry Ford Health System, Detroit, Michigan
  - Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina
  - The University of Toledo, Toledo, Ohio
  - The University of Oklahoma, Oklahoma City, Oklahoma
  - Lifespan Office of Research, Providence, Rhode Island
  - St. Joseph Hospital of Orange, Seattle, Washington